CLINICAL TRIAL: NCT03766217
Title: Bone Tissue Engineering With Dental Pulp Stem Cells for Alveolar Cleft Repair
Acronym: CLOSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Principal Investigator, Daniela Franco Bueno, Principal Investigator, Hospital Sirio-Libanes
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE47719215.5.0000.5461
Record Dates: First submitted 2018-11-29; First posted 2018-12-06 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Cleft Lip and Palate
MeSH Terms: conditions — Cleft Lip | interventions — Biocompatible Materials

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mesenchymal stem cells associated with biomaterials (Experimental): Mesenchymal stem cells obtained from autogenous deciduous dental pulp associated with biomaterials. The stem cells will be obtained by enzimatic digestion in GMP laboratory and will be seed into the biomaterial (hydroxyapatite/collagen).
  Interventions: Combination Product: Mesenchymal stem cells associated with biomaterials
- Iliac crest autogenous bone graft (Active Comparator): Autogenous bone will be obtained from iliac crest. The prepare of the receptor area will be the same in both arms and will follow current recommendations.
  Interventions: Combination Product: Iliac crest autogenous bone graft

INTERVENTIONS:
Combination Product: Mesenchymal stem cells associated with biomaterials — Deciduous dental pulp mesenchymal stem cells associated with hydroxyapatita/collagen.
  Arms: Mesenchymal stem cells associated with biomaterials
Combination Product: Iliac crest autogenous bone graft — Autogenous bone will be obtained from iliac crest.
  Arms: Iliac crest autogenous bone graft

SUMMARY:
Iliac crest autogenous bone graft is accepted as the most effective method for secondary alveolar cleft repair. However this method is associated with complications. As an alternative, mesenchymal stem cells associated with biomaterials have been used for the rehabilitation of the alveolar bone cleft of patients with cleft lip and palate. This is a RCT comparing mesenchymal stem cells obtained from autogenous deciduous dental pulp associated with biomaterials versus iliac crest autogenous bone graft for secondary alveolar cleft repair.

ELIGIBILITY:
Inclusion Criteria:

* non syndromic unilateral cleft lip and palate;
* age between 7 and 12 years;
* to have the jaw aligned and ready to receive the graft.

Exclusion Criteria:

* previous surgery to correct the alveolar cleft;
* have the canine erupted before grafting;
* incomplete orthodontic treatment;
* incomplete CT scan documentation.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Alveolar bone filling rate | 12 months
  Alveolar bone filling rate defined by the filling of at least 70% of the alveolar cleft area.
Serious adverse events | 12 months
  Serious adverse events resulting in death, life-threatening event, hospitalization, prolongation of existing hospitalization (for > 24 hours), persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions. Important medical event that may not result in death, be life threatening, or require hospitalization may be considered a serious adverse drug experience when, based upon medical judgment, it may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
  Frequency of participants experiencing at least one serious adverse event.

SECONDARY OUTCOMES:
Non serious adverse events | 15 days; 3, 6 and 12 months
  Frequency of participants experiencing at least one non serious adverse event
Bone Tissue Engineering With Dental Pulp Stem Cells for Alveolar Cleft Repair | Bone tissue engineering
Position of the canine tooth and formation of dental root | 12 months
  Position of the canine tooth and formation of dental root assessed by CT scan
Alveolar bone filling rate | 6 months
  Alveolar bone filling rate defined by the filling of at least 70% of the alveolar cleft area.
Serious adverse events | 15 days; 3 and 6 months
  Serious adverse events resulting in death, life-threatening event, hospitalization, prolongation of existing hospitalization (for > 24 hours), persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions. Important medical event that may not result in death, be life threatening, or require hospitalization may be considered a serious adverse drug experience when, based upon medical judgment, it may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
  Frequency of participants experiencing at least one serious adverse event.
Patient-reported outcome (PRO, including appearance, fuction and quality of life) | pre surgery and 12 months
  Assessed by CLEFT-Q, a self-report PRO instrument, tool answered independently patients themselves, without interpretation by the parent(s) or healthcare provider. The CLEFT-Q consists of 13 independently functioning domains (171 items) measuring appearance, facial function and quality of life. Each domain is composed of a series of items that together evaluate a unidimensional construct. A higher score means a better result (continuous outcome, measured by: mean)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sírio-Libanes, São Paulo, Brazil

REFERENCES:
- [Background] Tanikawa DYS, Pinheiro CCG, Almeida MCA, Oliveira CRGCM, Coudry RA, Rocha DL, Bueno DF. Deciduous Dental Pulp Stem Cells for Maxillary Alveolar Reconstruction in Cleft Lip and Palate Patients. Stem Cells Int. 2020 Mar 12;2020:6234167. doi: 10.1155/2020/6234167. eCollection 2020. PMID 32256610
- [Background] Pinheiro CCG, Leyendecker Junior A, Tanikawa DYS, Ferreira JRM, Jarrahy R, Bueno DF. Is There a Noninvasive Source of MSCs Isolated with GMP Methods with Better Osteogenic Potential? Stem Cells Int. 2019 Nov 6;2019:7951696. doi: 10.1155/2019/7951696. eCollection 2019. PMID 31781247